CLINICAL TRIAL: NCT06778941
Title: Etiology and Prognostic Analysis of Acute Liver Failure in Chinese Children: a Multi-center Bidirectional Observational Cohort Study
Brief Title: Etiology and Prognostic Analysis of Acute Liver Failure in Chinese Children
Acronym: EPOCH-ALF
Status: Not yet recruiting | Type: Observational
Sponsor: liyumei (Other)
Responsible Party: Sponsor-Investigator, liyumei, Professor, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Other Study IDs: 24K203-001; ChiCTR2400089260 (Registry Identifier: Chinese Clinical Trial Register (ChiCTR))
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Acute Liver Failure
MeSH Terms: conditions — Liver Failure, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Criteria for Diagnosing Pediatric Acute Liver Failure: This study is a multi-center, nationwide, dual-perspective, observational, open cohort study. It will recruit eligible hospitalized patients from the First Hospital of Jilin University and other participating institutions across the country for observation.

SUMMARY:
Research Background:

Pediatric acute liver failure (PALF) refers to the sudden onset of severe liver injury in children without known chronic liver disease, leading to multi-system organ dysfunction, with a mortality rate as high as 50%-70%. The etiology of PALF is complex and varied, including infections, metabolic disorders, and toxins. In developed countries, it is often caused by drug and toxin exposure, while in developing countries, viral infections are the primary cause. Additionally, 30%-50% of PALF cases have an unknown etiology, which increases the difficulty of treatment. Current treatment options include medical management, artificial liver support, and liver transplantation. Liver transplantation is the only proven effective treatment, but issues such as organ shortages and the timing of transplantation affect treatment outcomes. Improving diagnostic capabilities for the etiology and exploring optimal treatment strategies are of significant importance in enhancing the clinical success rate of PALF management.

Research Objective:

To explore the etiology and prognostic factors of pediatric acute liver failure (PALF), analyze the relationship between different causes of PALF and prognosis, and the relationship between different treatment modalities and prognosis. This study aims to investigate the correlation between etiology, treatment methods, and outcomes, providing scientific evidence to improve the precision in diagnosis and treatment of PALF and to enhance decision-making and timing judgments for liver transplantation.

DETAILED DESCRIPTION:
Data were organized and analyzed using WindRays statistical software. Quantitative data that followed a normal distribution were expressed as mean ± standard deviation (x ± s), and intergroup comparisons were performed using t-tests. For non-normally distributed quantitative data, median (interquartile range) [M (P25, P75)] was used, and intergroup comparisons were conducted using the Mann-Whitney U test. Qualitative data were presented as frequencies (n) and percentages (%), with intergroup comparisons made using χ² or Fisher's exact test. Multivariate logistic and Cox regression analyses were performed to adjust for potential confounding factors in the association between PALF etiology, treatment, and prognosis. Results were presented as odds ratios (ORs) with 95% confidence intervals (CIs). A multivariate-adjusted restricted cubic spline model was constructed to examine possible non-linear dose-response relationships between PALF etiology, treatment, and prognosis. Variables were selected using stepwise regression, lasso regression, and best subset regression. Risk scoring models were established using regression analysis, nomograms, scoring systems, decision trees, and machine learning algorithms. Sensitivity analyses were conducted using propensity score matching (PSM), regression analysis, and stratified analysis. The predictive efficacy of the model for PALF prognosis was evaluated using the area under the receiver operating characteristic (ROC) curve (AUC), with AUC ≥ 0.80 indicating good predictive value. Data with missing values less than 5% were deleted directly, and data with missing values between 5% and 20% were imputed using multiple imputation methods.

Handling of lost to follow-up: Multiple contact information and emergency contacts were collected at the beginning of the study to maintain regular communication with the patients and their guardians to reduce the risk of lost follow-up. If follow-up failed, multiple attempts were made to contact participants via phone, email, or other methods. Once lost to follow-up, multiple imputation methods were used to estimate missing data, and sensitivity analyses were conducted (if possible).

ELIGIBILITY:
Inclusion Criteria:

1. According to the diagnostic criteria for PALF, the following conditions must be met:

   ① Severe biochemical liver abnormalities occurring within 8 weeks;

   ② Coagulation disorders uncorrectable by vitamin K: if hepatic encephalopathy is present, prothrombin time (PT) > 15s or international normalized ratio (INR) > 1.5; regardless of the presence of hepatic encephalopathy, PT > 20s or INR > 2.0.
2. For patients who were admitted twice, only the information from the first hospitalization will be used.
3. Patients with a history of chronic liver disease (e.g., genetic metabolic factors, drug-induced factors) or biliary obstruction that led to the acute episode are categorized under acute liver failure.
4. The child's legal guardian has signed a written informed consent form.

Exclusion Criteria:

1. Age > 18 years;
2. Significant data missing (>10%);
3. The child's legal guardian refuses participation.

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Criteria for Diagnosing Pediatric Acute Liver Failure
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Discharge Status | At discharge (within 1 week)
  Cured:
  * Clinical symptoms such as bleeding tendency and hepatic encephalopathy disappear;
    * Jaundice resolves (TBil ≤ 2× upper limit of normal); ③ Liver function markers return to baseline; ④ PTA/INR normalizes.
  Improved:
  ① Significant improvement in clinical symptoms like bleeding, and disappearance of hepatic encephalopathy;
  * Significant improvement in jaundice, ascites, and other physical signs; ③ Liver function markers show marked improvement (TBIL < 5× upper limit of normal, PTA > 40% or INR < 1.5).
  Worsened:
  No improvement in symptoms or signs of liver failure, liver function deteriorates, and complications increase or worsen.
  Death or death within one week after withdrawal of treatment. Liver Transplantation.

IPD SHARING:
Plan to Share IPD: No
Due to privacy concerns and the sensitive nature of the data, we do not plan to share individual participant data with other researchers.